CLINICAL TRIAL: NCT07332767
Title: Myocardial Energetic Restoration in the Treatment of Obstructive Hypertrophic Cardiomyopathy
Acronym: MERIT HCM
Status: Not yet recruiting | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Wei Jun How, Cardiologist, University of Manchester
Other Study IDs: 367806
Record Dates: First submitted 2025-12-29; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Hypertrophic Cardiomyopathy (HCM)
Keywords: hypertrophic cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is the most common inherited heart condition, where the heart muscles can thicken to the point of obstructing blood flow out of the heart. This condition is associated with a chronic state of energy loss in the heart muscle.

Till more recently, a new class of medication (cardiac myosin inhibitors) have been introduced to directly target the heart muscle proteins (sarcomeres) to reduce the strength of contraction and relieve obstruction of blood flow out of the heart. While clinical trials have shown this class of medication significantly improves physical capacity and patient symptoms, it is still unclear, based on small scale published studies, where this improvement is achieved by restoring the fundamental energy balance within the heart.

Our research study aims to answer this question and prove mechanistic insights of the use of this class of medication in the HCM population with blood flow obstruction (otherwise known as obstructive HCM) by using a specialised non-invasive MRI technique which accurately measures the heart energy score (specifically known as the PCr/ATP ratio) in each participant. Our objective is to determine how a patient with obstructive HCM have their energy scores affected, and improve over time with this medication therapy. If positive, this finding could establish the use of PCr/ATP ratio as a crucial, objective biomarker for monitoring therapeutic response and informing personalised dosing strategies for patient in the future.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age and
* Have a confirmed diagnosis of oHCM that is not solely explained by abnormal loading conditions such as significant hypertension or valvular disease
* Qualify for mavacamten therapy by exhibiting a peak Left Ventricular Outflow Tract (LVOT) gradient of ≥ 50mmHg at rest or with provocation, New York Heart Association (NYHA) functional class II or III symptoms, and a baseline Left Ventricular Ejection Fraction (LVEF) of ≥ 55%

Exclusion Criteria:

* HCM phenocopies such as cardiac amyloidosis or Fabry's disease
* Undergone a septal reduction therapy (myectomy or ablation) within the preceding 6 months
* Any contraindications to mavacamten (e.g., baseline LVEF < 55%, pregnancy/breastfeeding)
* Inability to safely undergo a cardiac MRI, such as having non-compatible metal implants or severe claustrophobia

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort consists of adults diagnosed with symptomatic obstructive hypertrophic cardiomyopathy (oHCM) who are clinically eligible for and planning to initiate treatment with mavacamten.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-04-30 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Mean change in PCr/ATP ratio | 24 weeks
  The main goal is to determine if mavacamten therapy (cardiac myosin inhibitor) significantly improves the heart-muscle energy levels of patients with obstructive hypertrophic cardiomyopathy, as measured by the "energy score" (PCr/ATP) on a specialised MRI scan.

IPD SHARING:
Plan to Share IPD: Undecided